CLINICAL TRIAL: NCT02985047
Title: Brief Admission Skane: Can Brief Admission Replace General Admission for Individuals With Self-harm and Acute Risk of Suicide
Brief Title: Brief Admission Skane: Replacing General Admission for Individuals With Self-harm and Acute Risk of Suicide
Acronym: BAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Sofie Westling, MD, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/570
Record Dates: First submitted 2016-11-25; First posted 2016-12-07 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Self-Injurious Behavior; Suicidal Ideation; Suicide, Attempted; Borderline Personality Disorder; Emergency Services, Psychiatric
Keywords: Brief admission; admission; deliberate self-harm; self-harm
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide, Attempted; Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Admission (Experimental): Participants randomised to Brief admission (BA) will have the possibility of admitting themselves to hospital for a maximum duration of three consecutive days at a maximum frequency of three times per month. Apart from BA they have access to all psychiatric care that they would have if they had not participated in the study (including general admission to hospital).
  Interventions: Other: Brief Admission
- Control (No Intervention): Participants randomized to Treatment as Usual will receive no intervention from the study protocol, except the baseline assessments and repeated assessments administered on the same schedule as described above for the treatment group. They will not be given the evaluation measures that are specific to the intervention. Participants have access to all psychiatric care that they would have if they had not participated in the study (including general admission to hospital).

INTERVENTIONS:
Other: Brief Admission — Participants randomised to Brief admission (BA) will participate in a negotiation together with their out-patient clinician and a representative from the ward. The aim of the negotiation is to form an individualised contract defining how BA will work for them. After signing the contract, will have the possibility to admit themselves to hospital according to the procedure stated in the contract.
  Other Names: Brukarstyrd Inläggning (Swedish)
  Arms: Brief Admission

SUMMARY:
The purpose of the study is to test a standardized version of brief admission (BA) through randomized controlled trial (RCT). The main objective is to evaluate if BA can serve as a crisis management model for individuals with recurrent self-harm, including suicide attempts and at least three symptoms of Borderline Personality disorder. Participants will be allocated to BA + Treatment as Usual (TAU) or TAU.

DETAILED DESCRIPTION:
When individuals with recurrent self-harm and suicidal behaviour seek acute admission to hospital due to a crisis and associated increased suicidal ideation, recommendations for clinical care are still conflicting. The risk for iatrogenic effects of inpatient care are considerable, and long hospital admissions without a clear treatment structure may predict decompensation in functioning. This has resulted in a clinical practice of avoiding admission for individuals diagnosed with Borderline Personality Disorder (BPD).

Brief admission (BA) as an intervention has a longstanding history in the delivery of mental health services in the Netherlands. The core elements of brief admission were determined through consultation with Dutch researchers, interviews with individuals with experience, Dutch clinicians familiar with Brief Admission, and local guidelines from hospitals familiar with implementing this crisis management intervention. Core elements of the intervention were standardized into a protocol, and an educational manual was developed to train clinicians involved in the trial. An objectively rated fidelity measure was developed in order to ensure adherence.

ELIGIBILITY:
Inclusion Criteria:

* Current episodes of self-harm and/or recurrent suicidality.
* Fulfilling at least three criteria for borderline personality disorder.
* Admitted to psychiatric hospital for acute care for at least 7 days or presenting to the psychiatric emergency department at least 3 times during the last six months.

Exclusion Criteria:

* No regular contact with outpatient psychiatric services.
* Homelessness. Housing crises are outside the scope of this RCT.
* Medical disorder from other organs that significantly contributes to inclusion criteria (e.g. if self-harm only occurs during episodes of hypoglycemia in a diabetic patient).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Number of days with hospital admission | Change between the period from 12 month retrospectively to Baseline and the period from baseline to 12 months prospectively
  Number of days with Brief admission, general admission, forced (involuntary) admission

SECONDARY OUTCOMES:
Frequency of forced acts (e.g. restraints and forced medication) | Change between the period from 12 month retrospectively to Baseline and the period from baseline to 12 months prospectively
Individuals' Experiences of the intervention | Data collected at each Brief Admission during a period of 140 weeks. A Brief Admission is defined as a hospital admission according to the procedure defined in the Brief Admission Skane Standardised Protocol.
  Outcome from the questionnaires developed for the method: Individual's Experience Scale (IES)
Clinicians' Experiences of the intervention | Data collected at each Brief Admission during a period of 140 weeks. A Brief Admission is defined as a hospital admission according to the procedure defined in the Brief Admission Skane Standardised Protocol.
  Outcome from the questionnaires developed for the method: Clinician's Experience Scale (CES)
Frequency of all self-harming behaviours including suicide attempts | Change in frequency between baseline, 6 months and 12 months prospectively.
  Outcome from Five Self-Harm Behaviour Groupings Measure (5S-HM)
Severity of self-harming behaviours | Change in severity between baseline, 6 months and 12 months prospectively.
  Outcome from Five Self-Harm Behaviour Groupings Measure (5S-HM)
Level of functioning in activities of daily life | Change in ratings between baseline, 6 months and 12 months prospectively.
  The World Health Organization Disability Assessment Schedule II (WHODAS 2.0)
Ability to cope effectively with life stress | Change in ratings between baseline, 6 months and 12 months prospectively.
  The Brief COPE
Ability to regulate emotions | Change in ratings between baseline, 6 months and 12 months prospectively.
  The Difficulties in Emotion Regulation Scale
Global psychiatric symptoms | Change in ratings between baseline, 6 months and 12 months prospectively.
  Outcome from Clinical Global Impression Severity Scale
Satisfaction with health care | Change in ratings between baseline, 6 months and 12 months prospectively.
  Client Satisfaction Questionnaire (CSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westling, MD PhD, Principal Investigator — Region Skåne
Locations (1):
- Division of Psychiatry, Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Westling S, Daukantaite D, Liljedahl SI, Oh Y, Westrin A, Flyckt L, Helleman M. Effect of Brief Admission to Hospital by Self-referral for Individuals Who Self-harm and Are at Risk of Suicide: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195463. doi: 10.1001/jamanetworkopen.2019.5463. PMID 31173128
- [Derived] Helleman M, Lundh LG, Liljedahl SI, Daukantaite D, Westling S. Individuals' experiences with brief admission during the implementation of the brief admission skane RCT, a qualitative study. Nord J Psychiatry. 2018 Jul;72(5):380-386. doi: 10.1080/08039488.2018.1467966. Epub 2018 Apr 27. PMID 29703119
- [Derived] Liljedahl SI, Helleman M, Daukantaite D, Westrin A, Westling S. A standardized crisis management model for self-harming and suicidal individuals with three or more diagnostic criteria of borderline personality disorder: The Brief Admission Skane randomized controlled trial protocol (BASRCT). BMC Psychiatry. 2017 Jun 15;17(1):220. doi: 10.1186/s12888-017-1371-6. PMID 28619050

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT02985047/Prot_SAP_000.pdf